CLINICAL TRIAL: NCT06642103
Title: The Effect of Pain, Muscle Strength, Motor Imagery and Body Awareness on Function in Individuals With Chronic Lateral Epicondylitis
Brief Title: Pain, Muscle Strength, Motor Imagery, Body Awareness on Function and Individuals With Chronic Lateral Epicondylitis
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hasan Gerçek, Principle Investigator, KTO Karatay University
Other Study IDs: KaratayUH13
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to examine the effect of muscle strength, pain, motor imagery and body awareness on function in individuals with lateral epicondylitis. The main question it aims to answer is: Do pain, motor imagery, muscle strength and body awareness have an impact on function in individuals with lateral epicondylitis?

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of chronic LET by a physician and
* a pain score > 3 on a visual analog scale (VAS).

Exclusion Criteria:

* concomitant disorders of the wrist and forearm, such as elbow fracture or dislocation, and treatment with corticosteroid injections within the previous 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lateral epicondylitis
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Function | baseline
  Fuction will be evaluated with Patient-Rated Tennis Elbow Evaluation. The Patient-Rated Tennis Elbow Evaluation (PRTEE), is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis. The PRTEE allows patients to rate their levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales:
  Pain subscale - 5 items (0 = no pain, 10 = worst imaginable) Function subscale (0 = no difficulty, 10 = unable to do) Specific activities - 6 items Usual activities - 4 items

SECONDARY OUTCOMES:
Pain severity | Baseline
  The rest, activity and night pains of the participants will be evaluated with a 10 cm Visual Analog Scale before the treatment and at the end of the 4-week application. "0" means no pain, "10" means excruciating pain. Results will be recorded in cm.
Motor imagery | Baseline
  Motor imagery will be assessed through a left/right judgment task in which participants will need to recognize whether hand images correspond to their left or right side using the Recognise™ application (Neuro Orthopaedic Institute, Adelaide, Australia). For this test, participants will be seated comfortably in front of a table, with both elbows flexed at 90◦ and both index fingers placed on the bottom of the screen of an electronic tablet. Forty images of hands (20 on each side) in multiple postures, angles and skin colors will be randomly displayed in the center of the screen of the device. Participants will be given standard instructions to decide as quickly and accurately as possible whether each image is of the right or left hand by clicking on the 'left' (with left fingers) or 'right' (with right fingers) buttons shown at the bottom of the screen.
Grip strength | Baseline
  The maximal grip strength of the patients will be measured with a hydraulic hand dynamometer.
The Body Awareness | Baseline
  The Body Awareness Questionnaire will be used to assess body awareness. The questionnaire consists of 18 questions. Participants will be asked to score each statement on a scale ranging from 1 (1: Not true at all) to 7 (7: Completely true) and the total score will be obtained by summing the score given for each statement.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No